CLINICAL TRIAL: NCT03608280
Title: Evaluation of the Efficiency for Orbital Reconstruction After Defect of Bone Substance by Three-dimensional Printed Patient Specific Porous Titanium Implant in Comparison With Autologous Bone Graft
Brief Title: Efficiency of 3D-printed Implant Versus Autograft for Orbital Reconstruction (TOR-3D)
Acronym: TOR-3D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL18_0049; 2019-A02556-51 (Other: ANSM)
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Significant Bone Defect in the Orbit
Keywords: orbital reconstruction; 3D-printed patient specific porous titanium implant; autologous bone graft; medico-economic study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autograft (Active Comparator): Reconstructive surgery by autologous bone graft (bone autograft). It is the gold standard strategy.
  Interventions: Procedure: Bone autograft
- 3D implant (Experimental): Orbital reconstruction by 3D-printed porous titanium implant (PorousiTi®, laboratoire OBL/MATERIALISE).
  The device is a custom-made porous titanium implant processed by selective laser melting (SLM technique)
  Interventions: Procedure: Orbital reconstruction by 3D-printed porous titanium implant

INTERVENTIONS:
Procedure: Bone autograft — The principle of this surgery is based on the removal of a portion of the outer bone layer from the vault of the skull in order to have a flat and solid bone element (cortical bone), which can be carved freehand to better replace the defective bone wall.
  Arms: Autograft
Procedure: Orbital reconstruction by 3D-printed porous titanium implant — From data of a patient's CT-scan, it is possible to perform a "mirroring". The unaffected orbit is mirrored onto the affected orbit, via a virtual treatment planning, in order to rely on facial symmetry to virtually restore healthy anatomy. From this simulation, the implant is 3D-printed by Selective Laser Melted (SLM) technique using titanium powder. This technique enabling the creation of custom-made implants is called computer-aided design and computer-aided manufacturing (CAD-CAM).
  After sterilization, the implant is ready to be placed during a surgical procedure.
  Arms: 3D implant

SUMMARY:
Two scenarios may result in significant bone defect in the orbit: surgical oncology (meningioma, cancers of the upper aerodigestive tract) or severe trauma. This defect in the bone substance may affect the orbital floor, medial wall or lateral wall. These injuries can result in functional complications such as enophthalmos and diplopia, and an esthetic impact affecting the quality of life. The most frequent complication in orbital traumas is enophthalmos (10-20% according to publications).

The aim of bone substance reconstruction is to restore the volume and the internal shape of the orbit. The gold standard is autologous bone grafts. The surgery which usually lasts 2 to 3 hours depending on the number of walls involved, can lead to ophthalmological or esthetic complications. Its results are unsatisfactory, and the use of titanium implants would allow a reconstruction of the orbital volume more optimal than the autograft.

The development of computer-assisted techniques permitted implants evolution: initially peri-operatively preformed, today patient specific implant can be obtained from data of CT-scan. In cranioplasties, a randomized study showed better results at 12 months of these implants compared to the autograft. Their success rate is close to 100% with less than 5% of postoperative complication, while the rate used for cortical graft reconstructions is 20-25%.

Today, 3D printing of patient-specific porous titanium implants is possible. A study has shown that they allow a more accurate reconstruction compared to preformed implants. This innovation is available in France but it has a high cost (2,000 euros on average) and is currently not refunded. However, the use of this technology would reduce the operating time and the morbidity per- and post-operative, with functional and esthetic results superior to those obtained with bone autograft.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 to 90 years old
* Presenting a defect in the bone substance of an orbital wall (floor, lateral or medial): at least 6 months following a oncologic surgery (in particular meningioma or carcinoma of the upper aerodigestive tract) OR post-traumatic;
* With a defect of the unilateral orbital bone substance described as complex on the CT-scan: fracture in the posterior third of one walls; fracture extended to two walls (floor and lateral wall, or medial wall and orbital floor); comminutive fracture of at least one of the walls; fracture with more than half of one of the walls tipped over;
* Presenting an enophthalmos ≥ 3 mm OR an enophthalmos ≥ 2mm with diplopia;
* Patient with a programmed orbital reconstruction;
* For patients who have had oncologic surgery, validation of a multidisciplinary consultation meeting;
* Whose contralateral orbital anatomy is healthy (absence of : bone defect, diplopia, ptosis or other condition affecting aesthetics);
* Patient who gave its written informed consent to participate to the study;
* Affiliated to a social insurgence regime or similar.

Exclusion Criteria:

* Defect of bone substance extended to the upper and / or intermediate floors of the skull-base;
* For patients who have undergone oncologic surgery, patients with uncontrolled cancer proliferation;
* Defect of bone substance from the skull vault;
* Osteo-meningeal Breach;
* Patient whose understand the French questionnaire EQ-5D-3L;
* Follow up not possible during 18months (judgement of investigator)
* Patient with hypersensitivity to metallic materials;
* Major patient protected by the Law;
* Pregnant or breastfeeding woman

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incremental cost per quality-adjusted life-years (QALY) gained | 18 months
  QALY will be measured by EQ-5D-3L questionnaire. At 18 months post reconstruction, we can estimate most of the costs of surgery and its consequences.
  Incremental cost per quality-adjusted life-years (QALY) gained between patients with 3D-printed patient specific porous titanium implant or autologous bone graft for orbital reconstruction.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Groupement Hospitalier Sud Chirurgie maxillo-faciale, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: Undecided